CLINICAL TRIAL: NCT04897568
Title: Shared Decision Making in Rural Primary Care Lung Cancer Screening and Smoking Cessation
Acronym: SDM-LCS-SC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: High Plains Research Network (Network); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 19-1706.cc; P50CA244688 (NIH); NCI-2021-04394 (Other: CTRP)
Record Dates: First submitted 2021-03-03; First posted 2021-05-21 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Lung Cancer; Smoking Cessation
MeSH Terms: conditions — Lung Neoplasms; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: A type II effectiveness implementation hybrid trial will be conducted using a pre-post design to evaluate the effectiveness (co-primary outcomes of LCS and decision quality) and implementation at four rural clinics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will consist of each participant and clinic before the intervention (baseline, first 2 months).
- Patient decision aid (Active Comparator): The intervention group will consist of each participant and clinic once they move to the intervention phase (after the first 2 months).
  Interventions: Other: Patient decision aid

INTERVENTIONS:
Other: Patient decision aid — Each subject will receive an informational flyer describing lung cancer screening options and smoking cessation from a trained person on the medical staff at each clinic. Staff will lead a shared decision-making discussion with the patient.
  Other Names: Informational flyer
  Arms: Patient decision aid

SUMMARY:
The intervention is aimed to improve adherence to the lung cancer screening (LCS) guidelines and Centers for Medicare and Medicaid Services (CMS) coverage criteria to conduct shared decision-making (SDM) and provide smoking cessation services in rural primary care practices.

DETAILED DESCRIPTION:
The pilot intervention will engage no more than 300 patients using a pragmatic, pre-post design guided by an enhanced RE-AIM/PRISM framework. The primary goal of this intervention is to improve LCS practice by offering a formal SDM process and smoking cessation support aligned with the CMS coverage criteria. The investigators will conduct a type II effectiveness implementation hybrid trial using a pre-post design to evaluate the effectiveness (co-primary outcomes of LCS and decision quality) and implementation at four rural clinics. Space precludes discussion of pragmatic design features, but this study was designed to be pragmatic using the PRECIS-2 criteria and it scores highly on almost all PRECIS-2 dimensions.

Each clinic will recruit the minimum of 9 patients eligible to LCS (based on CMS guidelines) every 2 months for up to 8 months. The first period of 2 months is for baseline data, the second and every other period of 2 months is for intervention (pre-post design). Each patient will receive 2 surveys (one immediately after the doctor's visit and a second one a month later). The intervention will be in the form of patient decision aid (information flyer) the participant receives during a healthcare provider visit.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic to lung cancer symptoms
* Tobacco smoking history of 20+ pack-years
* Current smoker or quit within last 15 years

Exclusion Criteria:

- A patient that does not meet inclusion criteria

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Glasgow, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: clinic
Groups:
- Control (Pre-intervention): The control group will consist of each participant and clinic before the intervention (baseline, first 2 months).
- Patient Decision Aid (Post-intervention): The intervention group will consist of each participant and clinic once they move to the intervention phase (after the first 2 months, pre-post study design).
  Patient decision aid: Each subject will receive an informational flyer describing lung cancer screening options and smoking cessation from a trained person on the medical staff at each clinic. Staff will lead a shared decision-making discussion with the patient.
Period: Overall Study
Arm/Group | Control (Pre-intervention) | Patient Decision Aid (Post-intervention)
Started | 64; 3 clinic | 56; 3 clinic
Completed | 64; 3 clinic | 56; 3 clinic
Not Completed | 0; 0 clinic | 0; 0 clinic

BASELINE CHARACTERISTICS:
Population: Patients
Groups:
- Patient Decision Aid (Post-intervention): The intervention group will consist of each participant and clinic once they move to the intervention phase (pre-post design)
  Patient decision aid: Each subject will receive an informational flyer describing lung cancer screening options and smoking cessation from a trained person on the medical staff at each clinic. Staff will lead a shared decision-making discussion with the patient.
- Total: Total of all reporting groups
Arm/Group | Control (Pre-intervention) | Patient Decision Aid (Post-intervention) | Total
Number analyzed (Participants) | 64 | 54 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 42 | 94
  >=65 years | 12 | 12 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 28 | 61
  Male | 31 | 26 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 58 | 48 | 106
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants Who's Health Visit Adhered to the LCS Guidelines and CMS Coverage Criteria in Rural Primary Care Practices: Baseline Survey
Description: The adherence to the LCS guidelines and CMS coverage criteria to conduct SDM and provide smoking cessation services in rural primary care practices (is a latent variable) and will be measured as a composite measure using variables in a baseline survey administered immediately after healthcare provider's visit (baseline).
  A survey tool will be developed and used to count "Yes" response to the following survey questions:
  Were you given a decision aid during your last clinic visit/call? Was the clinic provider or staff able to go over the decision aid together with you during your last clinic visit/call? Were you recommended for a low-dose CAT scan by your provider during your last clinic visit/call?
Time Frame: Baseline
Measure: Number; unit: participants
Groups:
- Control: The control group will consist of each participant and clinic before the intervention (pre-intervention).
- Patient Decision Aid: The intervention group will consist of each participant and clinic once they move to the intervention phase (post-intervnetion).
  Patient decision aid: Each subject will receive an informational flyer describing lung cancer screening options and smoking cessation from a trained person on the medical staff at each clinic. Staff will lead a shared decision-making discussion with the patient.
Arm/Group | Control | Patient Decision Aid
Number analyzed (Participants) | 64 | 54
participants | 0 | 0

2. Primary Outcome: Count of Participants Who's Health Visit Adhered to the LCS Guidelines and CMS Coverage Criteria in Rural Primary Care Practices: Follow-up Survey
Description: The adherence to the LCS guidelines and CMS coverage criteria to conduct SDM and provide smoking cessation services in rural primary care practices (is a latent variable) and will be measured as a composite measure using variables in a baseline survey administered immediately after the healthcare provider's visit (follow-up).
  A survey tool will be developed and used to count "Yes" response to the following survey questions:
  Were you given a decision aid during your last clinic visit/call? Was the clinic provider or staff able to go over the decision aid together with you during your last clinic visit/call? Were you recommended for a low-dose computerized axial tomography (CAT) scan by your provider during your last clinic visit/call?
Time Frame: 1 month follow-up
Measure: Number; unit: participants
Groups:
- Patient Decision Aid: The intervention group will consist of each participant and clinic once they move to the intervention phase (stepped-wedge design: practices will be randomized into step 1, 2 or 3; for step 1: the intervention will start at 2 months, for step 2: the intervention will start at 4 months, for step 3: the intervention will start at 6 months).
  Patient decision aid: Each subject will receive an informational flyer describing lung cancer screening options and smoking cessation from a trained person on the medical staff at each clinic. Staff will lead a shared decision-making discussion with the patient.
Arm/Group | Control | Patient Decision Aid
Number analyzed (Participants) | 64 | 54
participants | 0 | 0

3. Secondary Outcome: Patient Knowledge About Lung Cancer
Description: Patient knowledge about lung cancer will be measured by overall knowledge score calculated from 15 survey questions previously used by Lau et al in their peer-reviewed manuscript published in the American Journal of Preventive Medicine titled Evaluation of a Personalized, Web-Based Decision Aid for Lung Cancer Screening. The level of knowledge will be assessed based on correct answers to 15 questions. The overall knowledge score will range from 0-15 where 0 is no correct answer (lowest knowledge) and 15 is all correct answers (highest knowledge).
  More correct answers indicate higher level of knowledge and higher score.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Patient Decision Aid
Number analyzed (Participants) | 64 | 54
score on a scale | 8.1 (2.3) | 8.5 (1.5)

4. Secondary Outcome: Patient Knowledge About Lung Cancer
Description: as for outcome 3
Time Frame: 1 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Patient Decision Aid
Number analyzed (Participants) | 64 | 54
score on a scale | 8.1 (2.3) | 8.5 (1.5)

ADVERSE EVENTS:
Time Frame: We did not collect adverse events data because our intervention involved reading a flyer.
Description: We did not collect adverse events data because our intervention involved reading a flyer.
Groups:
- Patient Decision Aid: The intervention group will consist of each participant and clinic once they move to the intervention phase (post-intervention).
  Patient decision aid: Each subject will receive an informational flyer describing lung cancer screening options and smoking cessation from a trained person on the medical staff at each clinic. Staff will lead a shared decision-making discussion with the patient.
Arm/Group | Control | Patient Decision Aid
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT04897568/Prot_SAP_001.pdf
  • Informed Consent Form: Postcard consent (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/68/NCT04897568/ICF_002.pdf